CLINICAL TRIAL: NCT01738984
Title: A Home Exercise Program for Women With Infants & Young Children
Acronym: MamaMove
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Klein Buendel, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9R42DA031402 (NIH)
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-03

CONDITIONS: MomZing Exercise Videos Online; Standard Exercise DVD
Keywords: exercise; video; DVD; mother; infant
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MomZing Web Program (Experimental): Features include selection one to three 10-minute videos demonstrating yoga, aerobics, and strengthening, specifically designed for mothers with infants 2 to 8 months of age. Women will sequence together videos personalized to their fitness level, preference for exercise type, and a choice to actively exercise with her baby or alone. Exercises with a baby will be tailored to the infant's weight and include interactions that promote cognitive development and mother-child bonding.
  Interventions: Behavioral: MomZing Web Program
- Standard exercise DVD (Experimental): Exercise DVD that demonstrates yoga or strengthening exercises a mother can perform with her infant.
  Interventions: Behavioral: Standard Exercise DVD

INTERVENTIONS:
Behavioral: MomZing Web Program — Online web platform that is accessed via a television connected to internet
  Arms: MomZing Web Program
Behavioral: Standard Exercise DVD — Standard exercise DVD that demonstrates exercises a women does with an infant.
  Arms: Standard exercise DVD

SUMMARY:
This Phase II Small Business Technology Transfer(STTR) project will develop and test the effectiveness of an interactive web program optimized for use on a Internet connected television(TV), titled Moms Exercising or (MomZing) that is designed specifically for women with infants 2-8 months old. Moms will select from a menu of 98, 10-minute exercise videos demonstrating yoga, aerobics, and strengthening exercises. They select and sequence together exercise videos personalized to their fitness level, form of exercise, and the choice to actively exercise with her baby or alone. The primary health goal of the MomZing Program is to increase home-based Moderate to Vigorous Physical Activity (MPVA) minutes per week in new mothers and to maintain their exercise increases over time as their baby grows.

The investigators hypothesize that women that use the MomZing Program will have greater increases in physical activity and fewer will return to cigarette smoking or alcohol use, compared to women who use a standard "mommy and me" exercise DVD.

DETAILED DESCRIPTION:
Becoming a mother is a significant transition in a woman's life, and while this is a positive experience for many, there can be significant decreases in healthful behaviors such as physical activity and increases in unhealthy behaviors including sleep deprivation, stress, and depressive symptoms. Increasing postpartum physical activity can have multiple health benefits including risk reduction for chronic diseases like diabetes and cardiovascular disease, and improvement in psychological health including decreased stress and depressive symptoms. Improvements in mental health outcomes can prevent substance use since psychological stress is a risk factor for substance use and abuse. The postpartum period also represents a critical period to prevent a return to substance use, including tobacco and alcohol.

This Small Business Technology Transfer(STTR)- Phase II project will develop and test an interactive web-enabled television program, titled Mothers Exercising or ("MomZing). Features include the ability to select one to five 10-minute videos demonstrating yoga, aerobics, and strengthening exercises for mothers with infants 2 to 8 months of age. Women will select and sequence together videos personalized to their fitness level, preference for exercise type, and the choice to actively exercise with her baby or alone. Exercises with a baby will be tailored to the infant's weight and include interactions that promote cognitive development and mother-child bonding. MomZing is designed for viewing on a television taking advantage of new technologies that allow viewers to watch streaming video (including movies) from the internet on a television. The television can also be connected to the internet via a web-enabled console such as an internet-connecting device.

The primary goal of the MomZing web-enabled Program is to increase home-based moderate-to-vigorous physical activity (MVPA) minutes per week in new mothers. Phase II activities will include: 1) programming the MomZing multimedia web enabled Program, a recruitment website, and online survey; 2) producing 98,10-minute video segments showing women exercising with or without an infant; 3) conducting iterative usability testing of the features and content of the Program; and, 4) conducting a randomized trial of the efficacy of the Program with 572 new mothers recruited from across the U.S. New mothers will be randomly assigned to receive either the MomZing web-enabled TV Program or a standard exercise DVD designed for new mothers. The primary outcome will be minutes per week of leisure-time moderate to vigorous physical activity measured at baseline, 4 and 12 weeks. Secondary outcomes include changes in fatigue, sleep, depressive symptoms, tobacco and alcohol use at 12 weeks. Process evaluation will also determine extent to which the technology is utilized (frequency of use and time per access) over 12 weeks in both conditions. We will investigate whether key demographic (i.e., weight of infant, number of children) physiological (i.e., body mass index), and lifestyle factors (sleep quality, fatigue) act as mediators or moderators of any change in physical activity.

The MomZing Program will allow Moms to tailor a range of exercise options to meet their needs and those of their infant. As their infant grows and progresses through different cognitive and developmental stages the Program can grow with them, allowing the Mom to change her preferences unlike any exercise multimedia(DVD or website) currently available on the market.

ELIGIBILITY:
Inclusion Criteria:

* woman aged 18-45 who has an infant 2-8 months old (who weighs 11-22 lbs)
* live in one of the 50 states in US
* have broadband, high speed wireless internet access at home
* have high definition, flat screen TV at home
* have DVD player at home
* sedentary (<30 minutes of exercise per week)
* BMI between 17-40
* healthy woman
* healthy infant
* likes to learn about new technology

Exclusion Criteria:

* woman has health problems: pregnant or planning to become pregnant in next 3 months, dizziness/loss of consciousness, bone/joint problems that would be made worse by exercise, cancer, coronary heart disease (chest pain),insulin dependent diabetic, exercise -induced asthma or other atherosclerotic cardiovascular diseases, on medication for heart condition/high blood pressure, doctor has limited the amount of physical exertion/exercising.
* Baby has health problems -a chronic illness/disorder that would prevent mother from holding or lifting him/her in her arms while exercising
* Woman cannot read/write English
* woman unable or unwilling to connect a device to her television at home to link it to her home's wireless network

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 499 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl L Albright, PhD, MPH, Principal Investigator — University of Hawaii
Locations (2):
- United States (2):
  - Cheryl Albright, PhD, MPH, Honolulu, Hawaii
  - University of Hawaii at Manoa, Honolulu, Hawaii

REFERENCES:
- See also: recruitment website — http://www.mamamove.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MomZing Web Program | Standard Exercise DVD
Started | 250 | 249
Completed | 186 | 210
Not Completed | 64 | 39
Not completed — Pregnancy | 4 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 59 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MomZing Web Program | Standard Exercise DVD | Total
Number analyzed (Participants) | 250 | 249 | 499
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (5.2) | 29.4 (5.3) | 29.8 (5.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 250 | 249 | 499
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 35 | 53
  Not Hispanic or Latino | 229 | 212 | 441
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 11 | 19
  Asian | 13 | 10 | 23
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 20 | 11 | 31
  White | 196 | 207 | 403
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 250 | 249 | 499
Minutes per week of moderate-to-vigorous of physical activity (MVPA min/wk) [Mean (Standard Deviation); unit: minutes per week] | 66.5 (99.7) | 85.8 (138.3) | 76.15 (119)
Number meeting goal of 150 moderate-to-vigorous min/week [Number; unit: participants] — For this outcome I wanted to report the percent of sample meeting goal of 150 minutes of moderate-to-vigorous physical activity per week and standard error - but drop downs below did not let me report percentage and SE - so listed just number for value
  participants | 45 | 71 | 116

OUTCOME MEASURES:

1. Primary Outcome: Minutes Per Week of Moderate-to-Vigorous Physical Activity (MPVA Min/wk) Assessed at 12 Weeks
Description: physical activity will be obtained via online surveys at the 12 week assessment point
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: MVPA minutes per week
Arm/Group | MomZing Web Program | Standard Exercise DVD
Number analyzed (Participants) | 186 | 210
MVPA minutes per week | 217.7 [202.9 to 233.1] | 203.2 [188.9 to 218.4]

2. Secondary Outcome: Number Who Returned to Smoking From Baseline and 12 Weeks
Description: change in smoking status between baseline and 12 week assessment will be collected via survey at baseline and at the 12 week survey
Time Frame: 12 weeks
Population: Number of participants who were not smoking at baseline but reported returned to smoking on 12 week survey.
Measure: Number; unit: participants
Arm/Group | MomZing Web Program | Standard Exercise DVD
Number analyzed (Participants) | 186 | 210
participants | 3 | 3

3. Other Pre Specified Outcome: Return to Drinking Between Baseline and 12 Weeks
Description: drinking status measured via online survey taken at baseline and 12 week
Time Frame: 12 weeks
Population: number of participants who never/rarely drank at baseline but reported drank 1 or more drink per week at 12 weeks.
Measure: Number; unit: participants
Arm/Group | MomZing Web Program | Standard Exercise DVD
Number analyzed (Participants) | 186 | 210
participants | 22 | 24

ADVERSE EVENTS:
Time Frame: Adverse event data collected at 4 and 12 weeks post baseline
Description: data reported by participants via online surveys
Arm/Group | MomZing Web Program | Standard Exercise DVD
Serious Adverse Events (participants affected / at risk) | 0/250 | 0/249
Other Adverse Events (participants affected / at risk) | 3/250 | 2/249
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MomZing Web Program (N=250) | Standard Exercise DVD (N=249)
Emergency appendectomy (Surgical and medical procedures) | 1 | 1
Broken foot bone (Musculoskeletal and connective tissue disorders) | 1 | 0
Torn meniscus (Musculoskeletal and connective tissue disorders) | 1 | 0
Surgery for herniated disk, pinched nerve (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No